CLINICAL TRIAL: NCT00433017
Title: 24-month Randomized, Double-masked, Controlled, Multicenter, Phase II Study Assessing Safety and Efficacy of Verteporfin Photodynamic Therapy Administered in Conjunction With Ranibizumab Versus Ranibizumab Monotherapy in Patients With Subfoveal Choroidal Neovascularization Secondary to AMD.
Brief Title: Verteporfin Photodynamic Therapy Administered in Conjunction With Ranibizumab in Patients With Subfoveal Choroidal Neovascularization Secondary to Age-related Macular Degeneration (AMD)
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Study was terminated based on the results of analyses performed as planned at Month 12.
Sponsor: Novartis (Industry)
Responsible Party: External Affairs, Novartis Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CBPD952A2309
Record Dates: First submitted 2007-02-08; First posted 2007-02-09 (Estimated); Results first posted 2011-02-04 (Estimated); Last update posted 2011-04-21 (Estimated); Status verified 2011-04

CONDITIONS: Macular Degeneration; Choroidal Neovascularization
Keywords: Age-related macular degeneration; AMD; Choroidal neovascularization; Verteporfin; Ranibizumab
MeSH Terms: conditions — Macular Degeneration; Choroidal Neovascularization | interventions — Verteporfin; Ranibizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Verteporfin + Ranibizumab (Experimental): Verteporfin (6 mg/m^2) photodynamic therapy (PDT) and ranibizumab (0.5 mg). Patients received three consecutive monthly ranibizumab injections starting on Day 1, and then as needed at intervals of at least 30 days based on retreatment criteria. These patients also received verteporfin PDT on Day 1 and then as needed from Month 3 at intervals of at least 90 days based on the retreatment criteria. From month 3 onward, retreatments were determined based on study-specific retreatment criteria that included retinal thickness by Optical Coherence Tomography (OCT), sub-retinal hemorrhage evaluated by ophthalmoscopic examination, visual acuity assessed using Early treatment Diabetic Retinopathy Study (ETDRS) visual acuity chart and CNV leakage assessed by fluorescein angiography (FA).
  Interventions: Drug: Verteporfin Photodynamic Therapy; Drug: Ranibizumab
- Ranibizumab Monotherapy (Active Comparator): Patients received three consecutive monthly ranibizumab injections starting on Day 1 and then as needed from Month 3 based on the retreatment criteria. These patients were also administered verteporfin placebo infusion with sham PDT on Day 1 and then as needed from Month 3 at intervals of at least 90 days based on the retreatment criteria. From month 3 onward, retreatments were determined based on study-specific retreatment criteria that included retinal thickness by Optical Coherence Tomography (OCT), sub-retinal hemorrhage evaluated by ophthalmoscopic examination, visual acuity assessed using Early treatment Diabetic Retinopathy Study (ETDRS) visual acuity chart and CNV leakage assessed by fluorescein angiography (FA).
  Interventions: Drug: Ranibizumab; Drug: Placebo

INTERVENTIONS:
Drug: Verteporfin Photodynamic Therapy — After a 10-minute intravenous infusion of verteporfin at a dose of 6 mg/m^2 body surface area, verteporfin was activated by light application of 50 J/cm^2 to the study eye, begun 15 minutes after the start of the infusion.
  Other Names: Visudyne
  Arms: Verteporfin + Ranibizumab
Drug: Ranibizumab — Ranibizumab 0.5 mg (0.05 mL of 10 mg/mL solution for injection) administered as an intravitreal injection
  Other Names: Lucentis
Drug: Placebo — As a placebo for verteporfin photodynamic therapy (for masking purposes), patients were administered a 10-minute intravenous infusion of 5% dextrose solution, followed by light application of 50 J/cm^2 to the study eye, begun 15 minutes after the start of infusion.
  Arms: Ranibizumab Monotherapy

SUMMARY:
This study will evaluate the effect of combination therapy with verteporfin photodynamic therapy and ranibizumab on visual acuity compared to ranibizumab monotherapy and the durability of response observed in patients with choroidal neovascularization secondary to age-related macular degeneration

ELIGIBILITY:
Inclusion Criteria:

* Subjects of either gender age 50 years or older
* Subfoveal choriodal neovascularization (CNV) due to age-related macular degeneration (AMD)

Exclusion Criteria:

* Choriodal neovascularization due to causes other than AMD
* Prior treatment for neovascular AMD in the study eye

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 255 (Actual)
Dates: Start 2007-05; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Chair — Novartis
Locations (12):
- Novartis Investigative site, Vienna, Austria
- Novartis Investigative site, Antwerp, Belgium
- Novartis Investigative site, Aalborg, Denmark
- Novartis Investigative site, Créteil, France
- Novartis Investigative site, Regensburg, Germany
- Novartis Investigative site, Budapest, Hungary
- Novartis Investigative site, Florence, Italy
- Novartis Investigative site, Rotterdam, Netherlands
- Novartis Investigative site, Warsaw, Poland
- Novartis Investigative site, Madrid, Spain
- Novartis Investigative site, Geneva, Switzerland
- Novartis Investigative site, Manchester, United Kingdom

REFERENCES:
- [Derived] Ritter M, Simader C, Bolz M, Deak GG, Mayr-Sponer U, Sayegh R, Kundi M, Schmidt-Erfurth UM. Intraretinal cysts are the most relevant prognostic biomarker in neovascular age-related macular degeneration independent of the therapeutic strategy. Br J Ophthalmol. 2014 Dec;98(12):1629-35. doi: 10.1136/bjophthalmol-2014-305186. Epub 2014 Jul 30. PMID 25079064
- [Derived] Larsen M, Schmidt-Erfurth U, Lanzetta P, Wolf S, Simader C, Tokaji E, Pilz S, Weisberger A; MONT BLANC Study Group. Verteporfin plus ranibizumab for choroidal neovascularization in age-related macular degeneration: twelve-month MONT BLANC study results. Ophthalmology. 2012 May;119(5):992-1000. doi: 10.1016/j.ophtha.2012.02.002. Epub 2012 Mar 17. PMID 22424834

RESULTS

PARTICIPANT FLOW:
Groups:
- Verteporfin + Ranibizumab: Patients received three consecutive monthly ranibizumab injections starting on Day 1, and then as needed at intervals of at least 30 days based on retreatment criteria. These patients also received verteporfin PDT on Day 1 and then as needed from Month 3 at intervals of at least 90 days based on the retreatment criteria. From month 3 onward, retreatments were determined based on study-specific retreatment criteria that included retinal thickness by Optical Coherence Tomography (OCT), sub-retinal hemorrhage evaluated by ophthalmoscopic examination, visual acuity assessed using Early treatment Diabetic Retinopathy Study (ETDRS) visual acuity chart and CNV leakage assessed by fluorescein angiography (FA).
- Ranibizumab: Patients received three consecutive monthly ranibizumab injections starting on Day 1 and then as needed from Month 3 based on the retreatment criteria. These patients were also administered verteporfin placebo infusion with sham PDT on Day 1 and then as needed from Month 3 at intervals of at least 90 days based on the retreatment criteria. From month 3 onward, retreatments were determined based on study-specific retreatment criteria that included retinal thickness by Optical Coherence Tomography (OCT), sub-retinal hemorrhage evaluated by ophthalmoscopic examination, visual acuity assessed using Early treatment Diabetic Retinopathy Study (ETDRS) visual acuity chart and CNV leakage assessed by fluorescein angiography (FA).
Period: Overall Study
Arm/Group | Verteporfin + Ranibizumab | Ranibizumab
Started | 122 | 133
Completed 12 Month Phase | 114 | 126
Completed | 26 | 32
Not Completed | 96 | 101
Not completed — Adverse Event | 5 | 3
Not completed — Withdrawal by Subject | 4 | 5
Not completed — Lost to Follow-up | 3 | 4
Not completed — Administrative problems | 80 | 86
Not completed — Protocol Violation | 1 | 0
Not completed — Death | 2 | 2
Not completed — Subject no longer requires study drug | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Verteporfin + Ranibizumab | Ranibizumab | Total
Number analyzed (Participants) | 122 | 133 | 255
Age Continuous [Mean (Standard Deviation); unit: years] | 76.8 (7.65) | 75.5 (7.44) | 76.1 (7.55)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 78 | 74 | 152
  Male | 44 | 59 | 103

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Best-corrected Visual Acuity (BCVA) at Month 12.
Description: BCVA score was based on the number of letters read correctly on the Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity chart assessed at a starting distance of 4 meters. An ETDRS visual acuity score of 85 is approximately 20/20. An increase in the VA score indicates improvement in visual acuity.
Time Frame: Baseline and Month 12
Population: Performed on the Full analysis set (FAS) using the Last Observation Carried Forward (LOCF) approach for imputing missing data. FAS consisted of all patients as randomized that received at least one application of study drug and had at least one post-baseline assessment for best corrected visual acuity in the study eye.
Measure: Mean (Standard Deviation); unit: Letters
Arm/Group | Verteporfin + Ranibizumab | Ranibizumab
Number analyzed (Participants) | 121 | 132
Letters
  Baseline | 54.6 (13.5) | 55.1 (12.3)
  Month 12 | 57.1 (18.3) | 59.4 (18.8)
  Change from Baseline | 2.5 (14.82) | 4.4 (15.92)

2. Primary Outcome: Percent of Participants With a Treatment-free Interval of at Least 3 Months Following the Month 2 Visit
Description: The number of patients with a ranibizumab treatment-free interval, ie, no active ranibizumab treatments for at least 3 months duration (at least 2 consecutive monthly visits), anytime following the Month 2 ranibizumab treatment. Only active ranibizumab treatments were considered.
Time Frame: Month 2 to Month 11
Population: Full analysis set. Includes number of participants in the treatment group with at least one visit assessment of re-treatment.
Measure: Number; unit: Percentage of Participants
Arm/Group | Verteporfin + Ranibizumab | Ranibizumab
Number analyzed (Participants) | 119 | 128
Percentage of Participants | 95.8 | 92.2

3. Secondary Outcome: Percentage of Patients With Fluorescein Leakage in the Study Eye at Month 12
Description: The proportion of patients with leakage of the study eye was assessed at the Central Reading Center (CRC) using Fluorescein angiography (FA).
Time Frame: Month 12
Population: The Full Analysis Set (FAS) based on observed data.
Measure: Number; unit: Percentage of participants
Arm/Group | Verteporfin + Ranibizumab | Ranibizumab
Number analyzed (Participants) | 97 | 115
Percentage of participants | 28.9 | 25.2

4. Secondary Outcome: Mean Change in Total Area of Leakage (Observed) of the Study Eye at Month 12
Description: Fluorescein angiography (FA) was used to assess the mean change of leakage of the study eye at the Central Reading Center (CRC). A negative change from baseline indicates improvement, ie, less leakage.
Time Frame: Baseline and Month 12
Population: Full analysis set based on observed data.
Measure: Mean (Standard Deviation); unit: mm^2
Arm/Group | Verteporfin + Ranibizumab | Ranibizumab
Number analyzed (Participants) | 92 | 107
mm^2
  Baseline | 7.4 (4.63) | 8.1 (5.82)
  Month 12 | 2.2 (4.88) | 2.0 (4.68)
  Change from Baseline | -5.3 (5.32) | -6.1 (6.44)

5. Secondary Outcome: Mean Change in Central Retinal Thickness of the Study Eye at Month 12
Description: Optical coherence tomography (OCT) was used to assess the mean change in retinal thickness of the study eye at the Central Reading Center (CRC). A negative change from baseline indicates improvement, ie, less thickness.
Time Frame: Baseline and Month 12
Population: Full analysis set, LOCF
Measure: Mean (Standard Deviation); unit: μm
Arm/Group | Verteporfin + Ranibizumab | Ranibizumab
Number analyzed (Participants) | 119 | 128
μm
  Baseline | 335.2 (94.7) | 339.8 (125.6)
  Month 12 | 219.9 (61.1) | 232.0 (54.5)
  Change from Baseline | -115.3 (98.7) | -107.7 (124.6)

ADVERSE EVENTS:
Time Frame: Includes cumulative data through 24 months.
Arm/Group | Verteporfin + Ranibizumab | Ranibizumab
Serious Adverse Events (participants affected / at risk) | 25/122 | 28/133
Other Adverse Events (participants affected / at risk) | 64/122 | 63/133
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Verteporfin + Ranibizumab (N=122) | Ranibizumab (N=133)
ANGINA PECTORIS (Cardiac disorders) | 1 | 1
ARRHYTHMIA (Cardiac disorders) | 0 | 1
ATRIAL FIBRILLATION (Cardiac disorders) | 1 | 0
ATRIAL FLUTTER (Cardiac disorders) | 0 | 1
CARDIAC FAILURE (Cardiac disorders) | 2 | 0
CARDIAC VALVE DISEASE (Cardiac disorders) | 1 | 0
CORONARY ARTERY DISEASE (Cardiac disorders) | 1 | 0
MYOCARDIAL INFARCTION (Cardiac disorders) | 2 | 0
MYOCARDIAL ISCHAEMIA (Cardiac disorders) | 1 | 0
CATARACT (Fellow eye) (Eye disorders) | 0 | 1
CATARACT (Study eye) (Eye disorders) | 0 | 2
CHORIORETINAL ATROPHY (Study eye) (Eye disorders) | 1 | 0
GLAUCOMA (Fellow eye) (Eye disorders) | 0 | 1
GLAUCOMA (Study eye) (Eye disorders) | 0 | 1
LAGOPHTHALMOS (Fellow eye) (Eye disorders) | 1 | 0
PARALYTIC LAGOPHTHALMOS (Study eye) (Eye disorders) | 0 | 1
RETINAL ARTERY OCCLUSION (Study eye) (Eye disorders) | 0 | 1
RETINAL CYST (Study eye) (Eye disorders) | 1 | 0
RETINAL DEGENERATION (Study eye) (Eye disorders) | 1 | 0
RETINAL OEDEMA (Study eye) (Eye disorders) | 1 | 0
ULCERATIVE KERATITIS (Fellow eye) (Eye disorders) | 1 | 0
VISUAL ACUITY REDUCED (Study eye) (Eye disorders) | 2 | 1
DIARRHOEA (Gastrointestinal disorders) | 0 | 1
GASTRITIS (Gastrointestinal disorders) | 0 | 1
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 | 0
HAEMORRHOIDS (Gastrointestinal disorders) | 1 | 0
HIATUS HERNIA (Gastrointestinal disorders) | 0 | 1
NAUSEA (Gastrointestinal disorders) | 0 | 1
SALIVARY GLAND CALCULUS (Gastrointestinal disorders) | 0 | 1
VISCEROPTOSIS (Gastrointestinal disorders) | 1 | 0
OEDEMA PERIPHERAL (General disorders) | 1 | 1
BILE DUCT STENOSIS (Hepatobiliary disorders) | 0 | 1
BILE DUCT STONE (Hepatobiliary disorders) | 0 | 1
ERYSIPELAS (Infections and infestations) | 1 | 0
LABYRINTHITIS (Infections and infestations) | 0 | 1
MASTOIDITIS (Infections and infestations) | 0 | 1
PNEUMONIA (Infections and infestations) | 1 | 0
SIALOADENITIS (Infections and infestations) | 0 | 1
WOUND INFECTION (Infections and infestations) | 1 | 0
CARTILAGE INJURY (Injury, poisoning and procedural complications) | 1 | 0
CONTUSION (Injury, poisoning and procedural complications) | 1 | 0
FALL (Injury, poisoning and procedural complications) | 4 | 2
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
HEAD INJURY (Injury, poisoning and procedural complications) | 0 | 1
HIP FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
JOINT DISLOCATION (Injury, poisoning and procedural complications) | 1 | 0
LUMBAR VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
MULTIPLE INJURIES (Injury, poisoning and procedural complications) | 0 | 1
UPPER LIMB FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
CARBOHYDRATE ANTIGEN 125 INCREASED (Investigations) | 1 | 0
HYPOKALAEMIA (Metabolism and nutrition disorders) | 0 | 1
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 1 | 0
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0
OSTEOPOROSIS (Musculoskeletal and connective tissue disorders) | 0 | 1
BLADDER NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
GENITAL NEOPLASM MALIGNANT FEMALE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
MEDIASTINUM NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
METASTASES TO PERITONEUM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
RENAL NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
SKIN CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
CAROTID ARTERY STENOSIS (Nervous system disorders) | 0 | 1
CEREBRAL ISCHAEMIA (Nervous system disorders) | 1 | 0
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 1 | 4
DIZZINESS (Nervous system disorders) | 0 | 2
FACIAL PARESIS (Nervous system disorders) | 0 | 1
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 0 | 1
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 1 | 0
SKIN ULCER (Skin and subcutaneous tissue disorders) | 0 | 1
AORTIC ANEURYSM (Vascular disorders) | 1 | 1
ARTERIAL STENOSIS LIMB (Vascular disorders) | 1 | 0
ARTERIAL THROMBOSIS LIMB (Vascular disorders) | 1 | 0
DEEP VEIN THROMBOSIS (Vascular disorders) | 0 | 1
ILIAC ARTERY OCCLUSION (Vascular disorders) | 1 | 0
ORTHOSTATIC HYPOTENSION (Vascular disorders) | 0 | 1
PERIPHERAL ARTERIAL OCCLUSIVE DISEASE (Vascular disorders) | 2 | 0
THROMBOSIS (Vascular disorders) | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Verteporfin + Ranibizumab (N=122) | Ranibizumab (N=133)
CONJUNCTIVAL HAEMORRHAGE (Study eye) (Eye disorders) | 4 | 10
EYE PAIN (Study eye) (Eye disorders) | 10 | 8
MACULAR DEGENERATION (Fellow eye) (Eye disorders) | 4 | 8
OCULAR HYPERAEMIA (Study eye) (Eye disorders) | 7 | 10
RETINAL HAEMORRHAGE (Study eye) (Eye disorders) | 7 | 5
BRONCHITIS (Infections and infestations) | 5 | 7
INFLUENZA (Infections and infestations) | 3 | 9
NASOPHARYNGITIS (Infections and infestations) | 18 | 15
INTRAOCULAR PRESSURE INCREASED (Study eye) (Investigations) | 11 | 8
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 8 | 3
HYPERTENSION (Vascular disorders) | 19 | 13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.